CLINICAL TRIAL: NCT04835246
Title: A Prospective, Single Centre Study Evaluating The Diagnostic Performance of Spectra IMDx System for The Detection of Gastric Cancer and Precancerous Lesions In Vivo
Brief Title: Evaluating Diagnostic Performance of Spectra IMDx System for Detection of Gastric Cancer and Precancerous Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Endofotonics Pte Ltd (Industry)
Collaborators: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EFCNX002
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Gastric Cancer; Gastric Precancerous Lesion
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spectra IMDx (Experimental): The physician will be asked to give a diagnosis of the lesion under White light endoscopy (WLE) firstly and the endoscopic diagnosis result will be recorded on case report form. Then the physician will introduce the probe of Spectra IMDx system to contact and assess the lesion. The Spectra IMDx system will detect the scattering light signal from the lesion and assess the risk of the lesion being high-grade intraepithelial neoplasia or gastric cancer, and display the result on the Spectra IMDx screen. The Spectra IMDx assessment will be recorded on case report form. Both the patient and doctor will be blinded from the results from Spectra IMDx system.
  After Spectra IMDx system examination, the physician takes biopsy sample(s) in suspected lesion for further histopathological diagnosis.
  Interventions: Device: Spectra IMDx system

INTERVENTIONS:
Device: Spectra IMDx system — The Spectra IMDx system is intended to be used in conjunction with conventional white light endoscopy in upper gastrointestinal endoscopic procedure to identify patients with high risk of developing and/or having gastric cancer and it is intended for use on patients above and equal to the age of 18.

SUMMARY:
The purpose of the study is to evaluate the diagnostic performance of a Raman spectroscopy analysis device - Spectra IMDx for the detection of gastric cancer and precancerous lesions in vivo.

DETAILED DESCRIPTION:
This is a prospective, single centre study to assess the diagnostic performance of Spectra IMDx system in detection of gastric cancer and precancerous lesions in subjects with suspected gastric intraepithelial neoplasia who are undergoing upper gastrointestinal endoscopic procedures.

The Spectra IMDx system comprises a laser system, a spectrometer, a computer with an analysis algorithm installed, and other ancillary parts. The Spectra IMDx system also comprises a Raman probe that can be connected with the main system. The Raman probe is an assembly of optical fibres and optical components arranged for maximal transmission of light energy. When in use, the laser system will emit a 785nm near infra-red laser that will be transmitted through the Raman probe to the distal end. When the laser is interrogated upon a tissue surface, the light energy is absorbed and reflected. The reflected energy is then collected from the distal end of the Raman probe, transmitted back to the main system, and passed through the spectrometer. The collected signal is then processed to obtain the clean Raman signal, which is then parsed through the analysis algorithm to evaluate its risk for cancer (high/low). Feedback will then be generated on the GUI in real time.

ELIGIBILITY:
Inclusion Criteria:

* The subject is older than 18 years of age.
* The subject is undergoing upper GI endoscopy for suspected intraepithelial neoplasia or gastric cancer lesions (less than 20mm)
* The subject must have personally signed and dated the patient informed consent form indicating that he/she has been informed of all pertinent aspects of the study.
* The subject must be willing and able to comply with all study procedures.

Exclusion Criteria:

* The subject has bleeding disorders, such as haemophilia, in whom biopsies are contraindicated.
* The subject shows presence of active gastrointestinal bleeding or coagulopathy precluding biopsies.
* The subject has rare gastric malignancies such as gastrointestinal stromal tumors (GISTs), lymphomas and neuroendocrine tumors （NETs）.
* The subject is pregnant.
* The subject with liver cirrhosis, impaired renal function, acute gastrointestinal (GI) bleeding, esophageal varices, jaundice, and GI post-surgery
* The subject with severe co-morbid illness, such as end-stage renal failure (ESRF), congestive cardiac failure (CCF), severe osteoarthritis (OA) and rheumatoid arthritis (RA) requiring long term non-steroidal anti-inflammatory drug (NSAID) therapy
* The subject has other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may interfere with the interpretation of study results and in the judgment of the investigator would make the subject unsuitable for entry into the study
* The subject on regular anti-coagulant prophylaxis such as warfarin must be able to undergo a five-day washout period before gastroscopy. The subject on aspirin, ticlopidine and clopidogrel must be able to undergo a one-week washout period before gastroscopy. The subject's physician or study co-investigator will exercise their clinical judgement to ensure subject's safety.
* The subject is unwilling or unable to provide signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Spectra IMDx system | During the procedure
  To assess the sensitivity of Spectra IMDx system for the detection of gastric cancer and precancerous lesions in vivo in the presence of using histological diagnosis as the gold standard.
  Diagnostic measurements will be assessed in this trial. Using the histopathological diagnosis as the gold standard, true positives (TPs), true negatives (TNs), false positives (FPs) and false negatives (FNs) can be obtained for both Spectra IMDx (IMDx) system.
  Sensitivity = TP/(TP + FN).

SECONDARY OUTCOMES:
Specificity of Spectra IMDx system | During the procedure
  To assess the specificity and accuracy of Spectra IMDx system for the detection of gastric cancer and precancerous lesions in vivo in the presence of using histological diagnosis as the gold standard.
  Specificity = TN/(TN + FP).
Accuracy of Spectra IMDx system | During the procedure
  To assess the accuracy of Spectra IMDx system for the detection of gastric cancer and precancerous lesions in vivo in the presence of using histological diagnosis as the gold standard.
  Accuracy = (TP + TN)/(TP + TN + FP + FN).

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhi Xu, MD, PhD, Principal Investigator — Zhongshan Hospital Xiamen University
Locations (1):
- Zhongshan Hospital Xiamen University, Xiamen, Fujian, China